CLINICAL TRIAL: NCT01367002
Title: Randomized Phase II Evaluation of Carboplatin/Paclitaxel With and Without Trastuzumab (Herceptin) in HER2/Neu+ Patients With Advance/Recurrent Uterine Serous Papillary Carcinoma
Brief Title: Evaluation of Carboplatin/Paclitaxel With and Without Trastuzumab (Herceptin) in Uterine Serous Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1012007786
Record Dates: First submitted 2011-05-26; First posted 2011-06-06 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Endometrial Cancer
Keywords: Uterine serous papillary carcinoma; Type II endometrial cancer; HER2/neu; Paclitaxel, Carboplatin, Trastuzumab
MeSH Terms: conditions — Endometrial Neoplasms | interventions — CP protocol; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carboplatin/Paclitaxel (Active Comparator): Chemotherapy
  Interventions: Drug: Carboplatin/Paclitaxel
- Trastuzumab (Experimental): Monoclonal antibody
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Carboplatin/Paclitaxel — Paclitaxel 175 mg/m2 will administered intravenously every 21 days for 6 cycles. Carboplatin AUC 5 will be administered intravenously every 21 days for 6 cycles. 100% of patients will receive Carboplatin/Paclitaxel.
  Other Names: Taxus brevifolia; cis-Diammine
  Arms: Carboplatin/Paclitaxel
Drug: Trastuzumab — Paclitaxel 175 mg/m2 will be administered intravenously every 21 days for 6 cycles. Carboplatin AUC 5 will be administered intravenously every 21 days for 6 cycles. On day 1, an 8 mg/kg loading dose of trastuzumab will be administered over a 90 minute period. Beginning on day 21, patients will receive 6mg/kg of trastuzumab, administered intravenously every 21 days and continued indefinitely every 21 days after 6 cycles of cytotoxic therapy are completed and until progression of the disease or prohibitive toxicities occur. 50% of patients will receive Carboplatin/Paclitaxel with the addition of Trastuzumab.
  Other Names: Herceptin
  Arms: Trastuzumab

SUMMARY:
The primary objective of this study is to estimate whether the addition of trastuzumab to paclitaxel and carboplatin chemotherapy improves progression free survival when compared to paclitaxel and carboplatin alone in Uterine Serous Papillary Carcinoma (USPC) patients overexpressing Her2/neu at 3+ level by immunohistochemistry (IHC)or positive by fluorescence in situ hybridization (FISH).

DETAILED DESCRIPTION:
The purpose of this study is to perform a randomized Phase II evaluation of Carboplatin/Paclitaxel with or without Trastuzumab (Herceptin) in patients with HER2/neu+ advanced stage/recurrent disease with an emphasis on determining the progression free survival in USPC patients and assessing immunologic markers predictive of trastuzumab response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced (stage III-IV) or recurrent histologically confirmed USPC with measurable disease.
* Patients must harbor a tumor HER2/neu+ based upon IHC staining score of 3+ or 2+ with confirmed gene amplification by FISH

Exclusion Criteria:

* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancers, significant history of cardiac disease, uncontrolled hypertension, unstable medical issue, brain leptomeningeal, prior therapy with trastuzumab, uncontrolled seizure disorder, seropositive for HIV, active hepatitis, hemorrhagic diathesis or requiring supplemental oxygen.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-06; Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D Santin, M.D., Principal Investigator — Yale University
Locations (20):
- United States (20):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - John Muir Clinical Research Center, Concord, California
  - Women's Cancer Research Foundation, Newport Beach, California
  - Penrose St. Francis Hospital, Colorado Springs, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - The University of Chicago Medicine, Chicago, Illinois
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - University of Maryland Medical Center, Silver Spring, Maryland
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Hilliard, Ohio
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Santin AD, Bellone S, Gokden M, Palmieri M, Dunn D, Agha J, Roman JJ, Hutchins L, Pecorelli S, O'Brien T, Cannon MJ, Parham GP. Overexpression of HER-2/neu in uterine serous papillary cancer. Clin Cancer Res. 2002 May;8(5):1271-9. PMID 12006548
- [Background] Santin AD, Bellone S, Siegel ER, Palmieri M, Thomas M, Cannon MJ, Kay HH, Roman JJ, Burnett A, Pecorelli S. Racial differences in the overexpression of epidermal growth factor type II receptor (HER2/neu): a major prognostic indicator in uterine serous papillary cancer. Am J Obstet Gynecol. 2005 Mar;192(3):813-8. doi: 10.1016/j.ajog.2004.10.605. PMID 15746676
- [Background] Santin AD, Bellone S, Van Stedum S, Bushen W, De Las Casas LE, Korourian S, Tian E, Roman JJ, Burnett A, Pecorelli S. Determination of HER2/neu status in uterine serous papillary carcinoma: Comparative analysis of immunohistochemistry and fluorescence in situ hybridization. Gynecol Oncol. 2005 Jul;98(1):24-30. doi: 10.1016/j.ygyno.2005.03.041. PMID 15894362
- [Background] Santin AD. Letter to the Editor referring to the manuscript entitled: "Phase II trial of trastuzumab in women with advanced or recurrent HER-positive endometrial carcinoma: a Gynecologic Oncology Group study" recently reported by Fleming et al., (Gynecol Oncol., 116;15-20;2010). Gynecol Oncol. 2010 Jul;118(1):95-6; author reply 96-7. doi: 10.1016/j.ygyno.2010.01.043. Epub 2010 Feb 20. No abstract available. PMID 20172595
- [Background] Schwartz PE. The management of serous papillary uterine cancer. Curr Opin Oncol. 2006 Sep;18(5):494-9. doi: 10.1097/01.cco.0000239890.36408.75. PMID 16894299
- [Background] Cirisano FD Jr, Robboy SJ, Dodge RK, Bentley RC, Krigman HR, Synan IS, Soper JT, Clarke-Pearson DL. The outcome of stage I-II clinically and surgically staged papillary serous and clear cell endometrial cancers when compared with endometrioid carcinoma. Gynecol Oncol. 2000 Apr;77(1):55-65. doi: 10.1006/gyno.2000.5737. PMID 10739691
- [Background] Goff BA, Kato D, Schmidt RA, Ek M, Ferry JA, Muntz HG, Cain JM, Tamimi HK, Figge DC, Greer BE. Uterine papillary serous carcinoma: patterns of metastatic spread. Gynecol Oncol. 1994 Sep;54(3):264-8. doi: 10.1006/gyno.1994.1208. PMID 8088602
- [Background] Randall ME, Filiaci VL, Muss H, Spirtos NM, Mannel RS, Fowler J, Thigpen JT, Benda JA; Gynecologic Oncology Group Study. Randomized phase III trial of whole-abdominal irradiation versus doxorubicin and cisplatin chemotherapy in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2006 Jan 1;24(1):36-44. doi: 10.1200/JCO.2004.00.7617. Epub 2005 Dec 5. PMID 16330675
- [Background] Burke TW, Gershenson DM, Morris M, Stringer CA, Levenback C, Tortolero-Luna G, Baker VV. Postoperative adjuvant cisplatin, doxorubicin, and cyclophosphamide (PAC) chemotherapy in women with high-risk endometrial carcinoma. Gynecol Oncol. 1994 Oct;55(1):47-50. doi: 10.1006/gyno.1994.1245. PMID 7959265
- [Background] Levenback C, Burke TW, Silva E, Morris M, Gershenson DM, Kavanagh JJ, Wharton JT. Uterine papillary serous carcinoma (UPSC) treated with cisplatin, doxorubicin, and cyclophosphamide (PAC). Gynecol Oncol. 1992 Sep;46(3):317-21. doi: 10.1016/0090-8258(92)90224-7. PMID 1526508
- [Background] Ball HG, Blessing JA, Lentz SS, Mutch DG. A phase II trial of paclitaxel in patients with advanced or recurrent adenocarcinoma of the endometrium: a Gynecologic Oncology Group study. Gynecol Oncol. 1996 Aug;62(2):278-81. doi: 10.1006/gyno.1996.0227. PMID 8751561
- [Background] Lincoln S, Blessing JA, Lee RB, Rocereto TF. Activity of paclitaxel as second-line chemotherapy in endometrial carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2003 Mar;88(3):277-81. doi: 10.1016/s0090-8258(02)00068-9. PMID 12648575
- [Background] Fleming GF, Brunetto VL, Cella D, Look KY, Reid GC, Munkarah AR, Kline R, Burger RA, Goodman A, Burks RT. Phase III trial of doxorubicin plus cisplatin with or without paclitaxel plus filgrastim in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2004 Jun 1;22(11):2159-66. doi: 10.1200/JCO.2004.07.184. PMID 15169803
- [Background] Ramondetta L, Burke TW, Levenback C, Bevers M, Bodurka-Bevers D, Gershenson DM. Treatment of uterine papillary serous carcinoma with paclitaxel. Gynecol Oncol. 2001 Jul;82(1):156-61. doi: 10.1006/gyno.2001.6211. PMID 11426978
- [Background] Creasman WT, Morrow CP, Bundy BN, Homesley HD, Graham JE, Heller PB. Surgical pathologic spread patterns of endometrial cancer. A Gynecologic Oncology Group Study. Cancer. 1987 Oct 15;60(8 Suppl):2035-41. doi: 10.1002/1097-0142(19901015)60:8+3.0.co;2-8. PMID 3652025
- [Background] Tymon-Rosario J, Siegel ER, Bellone S, Harold J, Adjei N, Zeybek B, Mauricio D, Altwerger G, Menderes G, Ratner E, Clark M, Andikyan V, Huang GS, Azodi M, Schwartz PE, Fader AN, Santin AD. Trastuzumab tolerability in the treatment of advanced (stage III-IV) or recurrent uterine serous carcinomas that overexpress HER2/neu. Gynecol Oncol. 2021 Oct;163(1):93-99. doi: 10.1016/j.ygyno.2021.07.033. Epub 2021 Aug 6. PMID 34372971
- [Result] Fader AN, Roque DM, Siegel E, Buza N, Hui P, Abdelghany O, Chambers SK, Secord AA, Havrilesky L, O'Malley DM, Backes F, Nevadunsky N, Edraki B, Pikaart D, Lowery W, ElSahwi KS, Celano P, Bellone S, Azodi M, Litkouhi B, Ratner E, Silasi DA, Schwartz PE, Santin AD. Randomized Phase II Trial of Carboplatin-Paclitaxel Versus Carboplatin-Paclitaxel-Trastuzumab in Uterine Serous Carcinomas That Overexpress Human Epidermal Growth Factor Receptor 2/neu. J Clin Oncol. 2018 Jul 10;36(20):2044-2051. doi: 10.1200/JCO.2017.76.5966. Epub 2018 Mar 27. PMID 29584549
- [Result] Fader AN, Roque DM, Siegel E, Buza N, Hui P, Abdelghany O, Chambers S, Secord AA, Havrilesky L, O'Malley DM, Backes FJ, Nevadunsky N, Edraki B, Pikaart D, Lowery W, ElSahwi K, Celano P, Bellone S, Azodi M, Litkouhi B, Ratner E, Silasi DA, Schwartz PE, Santin AD. Randomized Phase II Trial of Carboplatin-Paclitaxel Compared with Carboplatin-Paclitaxel-Trastuzumab in Advanced (Stage III-IV) or Recurrent Uterine Serous Carcinomas that Overexpress Her2/Neu (NCT01367002): Updated Overall Survival Analysis. Clin Cancer Res. 2020 Aug 1;26(15):3928-3935. doi: 10.1158/1078-0432.CCR-20-0953. Epub 2020 Jun 29. PMID 32601075

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel | Trastuzumab
Started | 29 | 32
Participants Receive Drug | 28 | 32
Participants Evaluable for PFS (PFS= Progression Free Survival) | 28 | 30
Completed | 28 | 30
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: Only those evaluable for PFS are included. Three were excluded due to: withdrawal of consent (n = 1) or failure to confirm HER2 positivity by fluorescence in situ hybridization (FISH) after 2+ immunohistochemistry (n = 2).
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin/Paclitaxel | Trastuzumab | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Median (Full Range); unit: years] | 73 [45 to 88] | 67 [57 to 85] | 69 [45 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 17 | 20 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58
Disease Status [Count of Participants; unit: Participants] — Uterine serous carcinoma (USC) advanced-stage primary or recurrent status
  Participants
    Advanced | 20 | 21 | 41
    Recurrent | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Differences Between Treatment Arms.
Description: Progression free survival differences between treatment arms.
Time Frame: 6 years
Population: Only patients eligible to be assessed for progression free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Paclitaxel | Trastuzumab
Number analyzed (Participants) | 28 | 30
months | 8.049 [7.129 to 9.692] | 12.945 [10.448 to 18.103]

2. Secondary Outcome: To Assess the Safety Profile of Trastuzumab in USPC Patients by CTCAE v4.0
Description: To assess the safety profile of trastuzumab in USPC patients by CTCAE v4.0. Presented are counts of those that experience any Serious Adverse Events or All Other Adverse Events.
Time Frame: 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel | Trastuzumab
Number analyzed (Participants) | 28 | 32
Participants
  Serious Adverse Events | 6 | 14
  All Other Adverse Events | 28 | 32

3. Secondary Outcome: To Assess Objective Response Rate (ORR)
Description: To assess objective response rate (ORR)
Time Frame: 6 years
Population: Among those with recurrent disease- see baseline characteristics table.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel | Trastuzumab
Number analyzed (Participants) | 8 | 9
Participants
  Complete Response (CR) | 2 | 1
  Partial Response (PR) | 4 | 3
  Stable Disease (SD) | 1 | 5
  Progressive Disease (PD) | 1 | 0

4. Secondary Outcome: To Assess Overall Survival (OS)
Description: To assess overall survival (OS), presented are the number of participants that survived through the duration of the study period.
Time Frame: 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel | Trastuzumab
Number analyzed (Participants) | 28 | 30
Participants | 7 | 9

ADVERSE EVENTS:
Time Frame: 30 days post treatment (treatment could last as long as 6 years)
Arm/Group | Carboplatin/Paclitaxel | Trastuzumab
All-Cause Mortality (participants affected / at risk) | 21/28 | 21/32
Serious Adverse Events (participants affected / at risk) | 6/28 | 14/32
Other Adverse Events (participants affected / at risk) | 28/28 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel (N=28) | Trastuzumab (N=32)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (2) | 0 (0)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (5)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fever (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel (N=28) | Trastuzumab (N=32)
Anemia (Blood and lymphatic system disorders) | 13 (33) | 16 (60)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (3) | 8 (28)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 2 (3) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 4 (6)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 3 (5)
Urinary tract infection (Infections and infestations) | 4 (5) | 6 (12)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (7)
Alkaline phosphatase increased (Investigations) | 4 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (5)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (2)
Cholesterol high (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 4 (7) | 9 (21)
Investigations - Other (Investigations) | 2 (3) | 2 (3)
Lymphocyte count decreased (Investigations) | 3 (4) | 2 (9)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 9 (38) | 11 (28)
Platelet count decreased (Investigations) | 6 (8) | 7 (10)
Weight gain (Investigations) | 0 (0) | 3 (9)
Weight loss (Investigations) | 1 (1) | 2 (3)
White blood cell decreased (Investigations) | 7 (36) | 6 (45)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (6) | 10 (16)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (6) | 8 (29)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 6 (8) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (9) | 5 (21)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (11) | 5 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 10 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (3) | 5 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (12) | 10 (16)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 8 (14)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (5) | 2 (3)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 6 (9)
Movements involuntary (Nervous system disorders) | 1 (1) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 2 (4)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (22) | 17 (24)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 4 (5) | 4 (4)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 5 (6) | 10 (11)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 6 (6) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 5 (8)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 2 (4)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (7) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (5) | 2 (2)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (3) | 1 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 10 (17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 10 (20)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (27) | 15 (30)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (7)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (6) | 7 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (2) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 5 (6) | 11 (22)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)
Vascular disorders - Other (Vascular disorders) | 1 (1) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Tinnitus (Vascular disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Vascular disorders) | 2 (2) | 1 (1)
Blurred vision (Eye disorders) | 2 (3) | 2 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 1 (2)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 16 (22)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (16) | 17 (26)
Diarrhea (Gastrointestinal disorders) | 5 (12) | 13 (30)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (3) | 6 (9)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 11 (16) | 18 (52)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 10 (17)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (7)
Chills (General disorders) | 1 (1) | 1 (2)
Fatigue (General disorders) | 17 (34) | 23 (62)
Fever (General disorders) | 2 (2) | 3 (5)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 2 (2) | 4 (6)
Pain (General disorders) | 2 (2) | 10 (19)
Edema limbs (General disorders) | 4 (5) | 7 (11)
Infusion related reaction (General disorders) | 0 (0) | 2 (2)
Localized edema (General disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT01367002/Prot_SAP_000.pdf